CLINICAL TRIAL: NCT02027610
Title: Newborn Vitamin A Supplementation, Gut Microbiota and Vaccine Response During the Second Year of Life in Bangladeshi Infants
Brief Title: Vitamin A, Stool Microbiota and Vaccine Response in Bangladeshi Infants
Status: Completed | Type: Observational
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); University of California, Davis (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: PR-13068
Record Dates: First submitted 2013-12-23; First posted 2014-01-06 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Vitamin A Deficiency
Keywords: Infant; Bangladesh; vitamin A; microbiota; vaccine; immunity
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Infant specimens containing DNA isolated from periferal blood mononuclear cells (PBMC) will be retained for future analyses. Maternal specimens containing DNA from cheek swabs will be retained for future analyses.
Oversight: Data Monitoring Committee: No

SUMMARY:
Vitamin A deficiency (VAD) increases the risk of death from infections in infants and young children. The World Health Organization (WHO) recommends high-dose vitamin A supplementation (VAS) from 6-59 months of age to reduce the risk of death in countries where VAD is common. Such countries include Bangladesh, where this study is being conducted. While providing VAS at 6 months is recommended, providing VAS at birth may also decrease the risk of death since newborn infants are also at risk of VAD. VAS presumably reduces infant mortality by improving the immune response to infection and immunization. Vitamin A particularly affects the development and function of T cells, which develop in the thymus and are a key component of the memory response to infection and immunization. Vitamin A is important for development of an important class of T cells, regulatory T-cells, in the intestine. Regulatory T-cells prevent over-reaction of the immune system to substances the immune system might otherwise treat as harmful such as food or the healthy bacteria in the intestine. VAD could disrupt the normal colonization of the infant's intestinal tract and cause a condition called "dysbiosis" where abnormal bacteria flourish and adversely affect the infant's immune system. Dysbiosis may disrupt the immune response to injectable and oral vaccines. VAS at birth may prevent dysbiosis and thus improve immune function, response to vaccines, and child survival. The investigators recently completed an intervention trial in Bangladeshi infants (NCT01583972) examining the effect of VAS at birth on immune function and response to vaccines administered from birth to 14 wk of age. The present study will recruit infants who completed NCT01583972 when they are from 12 to 24 m of age to determine if VAS at birth affects the responses to these same vaccines when they are measured during the second year of life. The investigators will examine the effect of VAS at birth on gut microbiota measured early in infancy and during the second year of life, and explore the association of the gut microbiota with vaccine response. Mothers of study infants will participate in the study because the breast milk oligosaccharide content strongly affects gut microbiota composition and the "secretor status" of the mother, which can be determined from maternal FUT2 genotype, strongly affects breast milk oligosaccharide content.

DETAILED DESCRIPTION:
Hypotheses and Specific Aims The investigators will test the hypotheses that VAS at birth will (1) improve production of new T cells at 1-2 yr of age; (2) improve T-cell memory responses at 1-2 yr of age to vaccines given early in infancy (birth - 14 wk); and (3) alter intestinal colonization early in infancy (6, 11 and 15 wk) and at 1-2 yr of age to increase Bifidobacterium and other healthy bacteria and decrease Proteobacteria and other harmful bacteria. Because the "secretor status" of the mother affects the carbohydrate content of the breastmilk, which can in turn affect Bifidobacterium growth in the infant gut, the "secretor status" of the mother will be determined. Furthermore these differences in composition of the intestinal bacteria will be associated with greater immunologic responses to oral and systemic vaccines.

Specific Aim 1: Determine if VAS or placebo at birth affect the blood concentration and thymic output of naïve T-cells at 1-2 yr of age. Specific Aim 2: Determine if VAS or placebo at birth affect T-cell mediated responses at 1-2 yr of age to vaccines given early in infancy, including serum and intestinal antibody levels, vaccine-specific proliferative responses by T cells and cytokine production by T cells. Specific Aim 3: Determine if VAS or placebo at birth affect the relative abundance of healthy intestinal bacteria and common harmful bacteria in the feces at 6, 11, and 15 wk of age and at 1-2 yr of age and determine if relative abundance of these bacteria correlates with vaccine responses shortly after vaccination (6, 11, 15 wk) and later in infancy (1-2 yr). As part of Aim 3 the "secretor status" genotype (FUT2 gene) of the mother will be determined from a cheek swab DNA sample.

ELIGIBILITY:
Inclusion Criteria:

* for infant: completion of NCT01583972
* for mother: mother of study infant

Exclusion Criteria:

* none

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The present study will recruit infants who completed NCT01583972 when they are from 12 to 24 months of age. Mothers of these infants will also be recruited for collection of DNA from a cheek swab.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Naïve T-cells in peripheral blood | measured once at 52 - 104 weeks of age
  The concentration of naïve T-cells in peripheral blood will be measured once at 52 - 104 wk of age by flow cytometric analysis.

SECONDARY OUTCOMES:
Thymic output of naïve T cells | measured once at 52 - 104 weeks of age
  The thymic output of naïve T cells will be measured once at 52 - 104 wk of age by T-cell receptor excision circle (TREC) levels in DNA purified from peripheral blood mononuclear cells (PBMC).
Immune response to vaccines | Measured once at 52 - 104 weeks of age
  The immune responses to vaccines, measured at 52 - 104 wk of age, include: (A) Serum immunoglobulin G (IgG) and immunoglobulin A (IgA) responses to oral polio virus vaccine (OPV; given at birth, 6 wk, 10 wk, 14 wk); (B) serum IgG response to tetanus toxoid vaccine (TT; given at 6, 10 and 14 wk) and (C) Hepatitis B virus vaccine (HBV; given at 6, 10 and 14 wk); (D) the IgA response to OPV in stool; the (E) proliferative and (F) cytokine response of peripheral blood cluster of differentiation 4 (CD4) T-cells to OPV, TT, HBV vaccines and to the tuberculosis vaccine (BCG; given at birth). Antibody responses will be measured by ELISA, T-cell proliferation by flow cytometric analysis after 6 days of culture with corresponding vaccine antigens, and cytokines will be measured in supernatant after 3 and 6 d of culture with the same antigens.
Change in the relative abundance of stool bacteria | 6, 10, 14 and 52-104 weeks of age
  The relative abundance of stool bacteria will be measured using DNA extracts at four time points (6, 10 and 14 wk, and at one point between 52 and 104 wk) using culture-independent, next generation sequencing (NGS) of bacterial populations, followed by quantitative PCR (QPCR) and Bifidobacterium-specific terminal restriction-fragment-length polymorphism (TRFLP.)
Serum Vitamin A status | measured once at 52-104 weeks of age
  Vitamin A status will be assessed by serum retinol or retinol binding protein (RBP4) at 52 - 104 wk of age.
Secretor status of the study infant's mother. | measured once when infant is 52 - 104 weeks of age
  The "secretor status" of the mother is determined by the FUT2 genotype. FUT2 is related to FUT1, the gene encoding fucosyltransferase 1, which determines the composition of specific glycans on erythrocytes that determine the ABO (or ABH) and Lewis blood group antigens. The activity of fucosyltransferase 2 (encoded by FUT2) causes the synthesis and secretion of these same glycans into breast milk and other secretions (e.g., saliva and other intestinal secretions).

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Stephensen, PhD, Principal Investigator — USDA, Western Human Nutrition Research Center
Locations (3):
- United States (2):
  - University of California, Davis, Davis, California
  - USDA Western Human Nutrition Research Center, Davis, California
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Derived] Ahmad SM, Huda MN, Raqib R, Qadri F, Alam MJ, Afsar MNA, Peerson JM, Tanumihardjo SA, Stephensen CB. High-Dose Neonatal Vitamin A Supplementation to Bangladeshi Infants Increases the Percentage of CCR9-Positive Treg Cells in Infants with Lower Birthweight in Early Infancy, and Decreases Plasma sCD14 Concentration and the Prevalence of Vitamin A Deficiency at Two Years of Age. J Nutr. 2020 Nov 19;150(11):3005-3012. doi: 10.1093/jn/nxaa260. PMID 32939553
- [Derived] Ahmad SM, Raqib R, Huda MN, Alam MJ, Monirujjaman M, Akhter T, Wagatsuma Y, Qadri F, Zerofsky MS, Stephensen CB. High-Dose Neonatal Vitamin A Supplementation Transiently Decreases Thymic Function in Early Infancy. J Nutr. 2020 Jan 1;150(1):176-183. doi: 10.1093/jn/nxz193. PMID 31504694
- [Derived] Huda MN, Ahmad SM, Kalanetra KM, Taft DH, Alam MJ, Khanam A, Raqib R, Underwood MA, Mills DA, Stephensen CB. Neonatal Vitamin A Supplementation and Vitamin A Status Are Associated with Gut Microbiome Composition in Bangladeshi Infants in Early Infancy and at 2 Years of Age. J Nutr. 2019 Jun 1;149(6):1075-1088. doi: 10.1093/jn/nxz034. PMID 31006815
- [Derived] Huda MN, Ahmad SM, Alam MJ, Khanam A, Kalanetra KM, Taft DH, Raqib R, Underwood MA, Mills DA, Stephensen CB. Bifidobacterium Abundance in Early Infancy and Vaccine Response at 2 Years of Age. Pediatrics. 2019 Feb;143(2):e20181489. doi: 10.1542/peds.2018-1489. PMID 30674610
- See also: International Centre for Diarrhoeal Disease Research, Bangladesh — http://www.icddrb.org/
- See also: United States Department of Agriculture, Western Human Nutrition Research Center — http://www.ars.usda.gov/Main/docs.htm?docid=11240